CLINICAL TRIAL: NCT05594719
Title: The Effect of Sun-like Spectrum With Different Spectrum Composition on Retinal Blood Flow in School Students: a Randomized Controlled Trial
Brief Title: The Effect of Sun-like Spectrum With Different Spectrum Composition on Retinal Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YFZXLDX20220801
Record Dates: First submitted 2022-10-01; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Myopia
Keywords: myopia; retinal blood flow; accommodative micro-fluctuation; artificial lighting
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: The participants were randomly divided into the following three groups:
  1. Sun-like spectrum, color temperature of 5000K, shorter-wavelength dominant;
  2. Sun-like spectrum, color temperature of 5000K, wavelength proportion similar to the sunlight;
  3. Sun-like spectrum, color temperature of 5000K, longer-wavelength dominant.
Who Masked: Participant
Masking Description: The participants were randomly divided into three groups without knowing the type of light
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light group 1 (Experimental): Sun-like spectrum, color temperature of 5000K, shorter-wavelength dominant;
  Interventions: Device: Shorter-wavelength dominant light
- Light group 2 (Placebo Comparator): Sun-like spectrum, color temperature of 5000K, wavelength proportion similar to the sunlight
  Interventions: Device: Light similar to the solar spectrum proportion
- Light group 3 (Experimental): Sun-like spectrum, color temperature of 5000K, longer-wavelength dominant.
  Interventions: Device: Shorter-wavelength dominant light; Device: Longer-wavelength dominant light

INTERVENTIONS:
Device: Shorter-wavelength dominant light — Shorter-wavelength dominant light
  Arms: Light group 1; Light group 3
Device: Light similar to the solar spectrum proportion — Light similar to the solar spectrum proportion with no specific wavelength dominant
  Arms: Light group 2
Device: Longer-wavelength dominant light — Longer-wavelength dominant light
  Arms: Light group 3

SUMMARY:
In 2020, the overall myopia rate among children and adolescents was 52.7% in China. The COVID-19 pandemic has increased students' time of indoor eye-using, and it showed that the light exposure intensity of myopic students is lower than that of non-myopia students. Studies have found that in addition to exposure to light intensity, the occurrence and development of myopia is also related to the color temperature and wavelength band of light. The sun-like spectrum refers to the spectrum with continuous wavelength bands. Animal experiments suggest that sun-like artificial lighting can prevent myopia, but the relationship between sun-like artificial lighting with different color temperatures and myopia is unknown. Clinical trials suggest that artificial lighting with a sun-like spectrum can delay fundus blood flow decline. One hypothesis is that reduced choroidal blood flow leads to scleral hypoxia and promotes the development of myopia. This study aims at comparing the effects of sun-like spectrum artificial lighting with different dominant wavelengths on the human eye, and providing clues for the prevention and control of myopia.

DETAILED DESCRIPTION:
In 2018, eight departments including the Ministry of Education jointly issued the Implementation Plan for Comprehensive Prevention and Control of Myopia in Children and Adolescents. As of 2020, the overall myopia rate among children and adolescents was 52.7% in China. The COVID-19 pandemic has increased students' time of indoor eye-using, and it showed that the light exposure intensity of myopic students is lower than that of non-myopia students. Studies have found that in addition to exposure to light intensity, the occurrence and development of myopia is also related to the color temperature and wavelength band of light. Animal experiments showed that the bandwidth of light had a significant effect on the emmetropia of the eye, and white light can promote emmetropia more than monochromatic light; longer-wavelength light and shorter-wavelength light can promote and inhibit the development of myopia through hyperopia and myopic defocus, respectively. At present, the artificial lighting methods on the market are mainly light emitting diode (LED), whose light spectrum is discontinuous. With the advancement of related research and lighting technology, multiple LED emission peaks and "sun-like spectrum" desk lamps have gradually appeared. The sun-like spectrum refers to the spectrum with continuous wavelength bands. Animal experiments suggest that sun-like artificial lighting can prevent myopia, but the relationship between sun-like artificial lighting with different color temperatures and myopia is unknown. Clinical trials suggest that artificial lighting with a sun-like spectrum can delay fundus blood flow decline. Fundus blood flow is sensitive to myopia stimuli, and is a short-term effect indicator of the relationship between light environment and myopia. One hypothesis is that reduced choroidal blood flow leads to scleral hypoxia and promotes the development of myopia. Therefore, in this study fundus blood flow was selected as the main research indicator, aiming to compare the effects of sun-like spectrum artificial lighting with different dominant wavelengths on the human eye, and provide clues for the prevention and control of myopia.

ELIGIBILITY:
Inclusion Criteria:

* School students aged from 7 to 15, regardless of sex or gender;
* Diopter between -2.0D and 3.0D, and astigmatism not exceed 0.75D;
* No organic disease and in good general condition;
* Have obtained the consent of their parents or guardians, and can cooperate.

Exclusion Criteria:

* Suffering from amblyopia, strabismus, color weakness, congenital cataract, glaucoma and other eye diseases;
* Other circumstances judged by the investigator to be unsuitable to participate in the research.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Retinal blood flow density after reading | At the timepoint after reading for 1 hour
  Data werevcollected from Optovue AngioVue OCT (macular blood data collected), dominant eye examined

SECONDARY OUTCOMES:
Accommodation ability after reading | At the timepoint after reading for 1 hour
  Data were collected from AcomoREF2 (AMF mode, record distance and high-frequency component), for the dominant eye. And the Accommodative response value was documented for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangui He, PhD, Principal Investigator — Shanghai Eye Hospital
Locations (2):
- China (2):
  - Xiangui He, Shanghai, Shanghai Municipality
  - Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirhajianmoghadam H, Pina A, Ostrin LA. Objective and Subjective Behavioral Measures in Myopic and Non-Myopic Children During the COVID-19 Pandemic. Transl Vis Sci Technol. 2021 Sep 1;10(11):4. doi: 10.1167/tvst.10.11.4. PMID 34473223
- [Background] Muralidharan AR, Lanca C, Biswas S, Barathi VA, Wan Yu Shermaine L, Seang-Mei S, Milea D, Najjar RP. Light and myopia: from epidemiological studies to neurobiological mechanisms. Ther Adv Ophthalmol. 2021 Dec 19;13:25158414211059246. doi: 10.1177/25158414211059246. eCollection 2021 Jan-Dec. PMID 34988370
- [Background] Rucker F. Monochromatic and white light and the regulation of eye growth. Exp Eye Res. 2019 Jul;184:172-182. doi: 10.1016/j.exer.2019.04.020. Epub 2019 Apr 21. PMID 31018118
- [Background] Baeza Moyano D, González-Lezcano RA. Pandemic of Childhood Myopia. Could New Indoor LED Lighting Be Part of the Solution? Energies. 2021;14(13):3827. doi:10.3390/en14133827
- [Background] 陈军, 陈友三, 王菁菁, et al. 类太阳光谱LED照明对儿童青少年视网膜血流灌注影响的随机对照临床试验. zgxxws. 2022;43(3):338-340. doi:10.16835/j.cnki.1000-9817.2022.03.005
- [Background] Liu Y, Wang L, Xu Y, Pang Z, Mu G. The influence of the choroid on the onset and development of myopia: from perspectives of choroidal thickness and blood flow. Acta Ophthalmol. 2021 Nov;99(7):730-738. doi: 10.1111/aos.14773. Epub 2021 Feb 7. PMID 33550704